CLINICAL TRIAL: NCT01384253
Title: Phase I Trial of Intraperitoneal ²¹²Pb-TCMC-Trastuzumab for HER-2 Expressing Malignancy
Brief Title: Safety Study of ²¹²Pb-TCMC-Trastuzumab Radio Immunotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orano Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AREVAMED01
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Breast Neoplasms; Peritoneal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms
Keywords: HER2+; HER-2 positive; intraperitoneal; intra-abdominal; Lead 212; Radio Immunotherapy; Alpha particle; Antibodies; Immunoglobulins; Antibodies, Monoclonal; Immunologic Factors; Physiological Effects of Drugs; Pharmacologic Actions; RIT
MeSH Terms: conditions — Breast Neoplasms; Peritoneal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I: Dose escalation (Experimental): In preparation for the study, patients screened and eligible will have a peritoneal catheter placed and the evening prior to the injection of the labeled antibody will receive furosemide. Herceptin will be administered IV followed by a single IP infusion of ²¹²Pb-TCMC-Trastuzumab. Serial sampling of blood, urine, and dosimetry will be performed following treatment to determine the toxicity, pharmacokinetics, immunogenicity, and antitumor effects.
  Interventions: Other: ²¹²Pb-TCMC-Trastuzumab; Biological: trastuzumab

INTERVENTIONS:
Other: ²¹²Pb-TCMC-Trastuzumab — The starting dose level will be 200 μCi/m² of ²¹²Pb-TCMC-Trastuzumab. Three to six patients will be treated at each dose level, and dose escalation will proceed if no more than 1 out of 6 patients in a cohort experiences dose limiting toxicity. Six patients will be treated at the maximum tolerated dose.
Biological: trastuzumab — 4 mg/kg.
  Other Names: Herceptin

SUMMARY:
Monoclonal antibodies can transport and deliver radioactive elements capable of releasing sufficient amounts of energy to destroy tumor cells. In this clinical trial, we will study alpha particle radio immunotherapy using lead-212 (²¹²Pb), an isotope with a short path length targeted to malignant cells by the trastuzumab antibody, as a potential treatment for metastatic diseases.

This Phase I trial is designed to determine the toxicity profile of ²¹²Pb-TCMC-Trastuzumab, its dose-limiting toxicities, and its anti-tumor effects in patients with HER-2 positive intraperitoneal cancers.

ELIGIBILITY:
Inclusion Criteria:

1. At least 19 years of age.
2. Life expectancy is greater than three months.
3. Female subjects of child-bearing potential must have negative serum pregnancy test.
4. If not surgically sterile, male and female patients of child-bearing potential must use double barrier contraception (e.g., hormonal; intrauterine device; barrier).
5. Patients with HER-2 expressing tumors (e.g., ovarian, pancreatic, colon, gastric, endometrial, or breast) with measurable or non-measurable disease for which no standard therapy is available.
6. HER-2 amplification by fluorescent in situ hybridization or HER-2 score of at least at least 1+ by Immunohistochemistry in more than 10% of the cells. Alternatively, HER-2 serum levels greater than 15ng/mL by ELISA.
7. Disease must be predominantly intra-abdominal and should include documented peritoneal studding or positive peritoneal washings.
8. Able and willing to sign an informed consent form.

Exclusion Criteria:

1. ECOG performance status greater than 3.
2. Any serious active disease or co-morbid condition that, in the opinion of the investigator, may interfere with the safety or the compliance with the study.
3. Poor bone marrow reserve as defined by absolute neutrophil count less than 1.5 x 10³/cmm or platelets less than 100 x 10³/cmm within two weeks prior to initiation of treatment.
4. Liver only metastases.
5. Poor organ function as defined by one of the following:

   * Total bilirubin greater than 1.5 upper limits of normal (ULN)
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) greater than 2.5 ULN or greater than 5 ULN in case of documented liver metastasis
   * Serum creatinine greater than ULN, except if calculated creatinine clearance greater than 60 mL/min
   * Urine Protein/Creatinine Ratio greater than 1 on morning spot urinalysis or proteinuria greater than 500 mg/24 h
6. Breast-feeding woman.
7. No resolution of all specific toxicities (excluding alopecia) related to any prior anticancer therapy to Grade 2 according to the National Cancer Institute common terminology criteria for adverse events (NCI CTCAE) v.4.03 or nausea and vomiting to Grade 3 and uncontrolled with anti-emetics.
8. Wash out period of less than three weeks from previous anti-tumor therapy or any investigational treatment (and less than six weeks in case of prior nitroso-urea and or mitomycin C treatment) of scheduled date of administration.
9. Wash out period of less than one week from last palliative dose of radiotherapy.
10. Any other severe underlying medical conditions that could impair the ability to participate in the study or the interpretation of its results related to the investigational product such as:

    * Patients with abnormal cardiac function defined by a left ventricular ejection fraction (LVEF) less than 50% by echocardiogram (ECHO) or multi gated acquisition (MUGA) scan
    * Patients with previous history of acute cardiac failure
11. Clinical symptoms of bowel obstruction, evidence of rectosigmoid bowel involvement on exam, or transmural bowel wall involvement on computed tomography (CT) or magnetic resonance imaging (MRI).
12. Prior whole abdomen radiation therapy exceeding 4Gy, intraperitoneal radionuclide therapy, bone marrow transplant, or stem cell transplant.
13. History of Human Immunodeficiency Virus (HIV) antibody by enzyme-linked immunosorbent assay (ELISA) or negative by Western blot (if ELISA is positive) or hepatitis B surface antigen (HBsAg) because of the potential for added toxicity from the radiolabeled antibody among patients infected with these viruses.
14. Detectable human anti-human antibody (HAHA) if there is any history of monoclonal antibody exposure.
15. Iodine allergy if the patient is unwilling to accept radiation to the thyroid from uptake of radionuclide without blocking.
16. Allergy to furosemide if the patient is unwilling to accept radiation risk without these agents and alternative is not feasible.
17. History of cumulative anthracycline therapy exceeding 200 mg/m² for doxorubicin or comparable low dose of other anthracyclines.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-07; Primary Completion 2015-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: To measure the number of participants who experience adverse events after intraperitoneal (IP) administration of ²¹²Pb-TCMC-Trastuzumab. | Assessed periodically during study treatment follow-up, up to five years.
  Adverse events considered dose limiting toxicity:
  * Grade 3 elevations of ALP, bilirubin, ALT, or AST lasting ≥7 days
  * Grade 3 elevations of serum creatinine within 6 weeks of treatment
  * Grade 2 elevations of serum creatinine lasting ≥7 days that occur after 6 weeks
  * Grade 3 proteinuria
  * Any other Grade 3 or 4 non-hematologic toxicity
  * Grade 4 neutropenia lasting ≥7 days or febrile neutropenia of any duration
  * Grade 3 thrombocytopenia that fails to recover to ≤ Grade 2 at 6 weeks
  * Grade 4 thrombocytopenia lasting ≥7 days or thrombocytopenia accompanied by bleeding

SECONDARY OUTCOMES:
Immunogenicity: To characterize the human immune response against ²¹²Pb-TCMC-Trastuzumab given via IP infusion. | Assessed at six weeks visit
Anti-tumor effects: To monitor for anti-tumor effects as assessed by physical examination, radiographic imaging, and tumor marker studies. | Assessed after six and twelve weeks, and then at twelve-week intervals until progression.
Pharmacokinetics: To determine the plasma pharmacokinetics and assess the extent of exit of radioactivity from the peritoneal cavity by γ-camera imaging. | Up to 3 days post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Ruby F Meredith, M.D., Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University Of Alabama at Birmingham, Birmingham, Alabama
  - UCSD Moores Cancer Center, San Diego, California

REFERENCES:
- [Background] Meredith RF, Torgue J, Azure MT, Shen S, Saddekni S, Banaga E, Carlise R, Bunch P, Yoder D, Alvarez R. Pharmacokinetics and imaging of 212Pb-TCMC-trastuzumab after intraperitoneal administration in ovarian cancer patients. Cancer Biother Radiopharm. 2014 Feb;29(1):12-7. doi: 10.1089/cbr.2013.1531. Epub 2013 Nov 14. PMID 24229395
- [Background] Meredith R, Torgue J, Shen S, Fisher DR, Banaga E, Bunch P, Morgan D, Fan J, Straughn JM Jr. Dose escalation and dosimetry of first-in-human alpha radioimmunotherapy with 212Pb-TCMC-trastuzumab. J Nucl Med. 2014 Oct;55(10):1636-42. doi: 10.2967/jnumed.114.143842. Epub 2014 Aug 25. PMID 25157044
- See also: University of Alabama at Birmingham Department of Oncology Clinical Research — http://www.uab.edu/radonc/clinical-research.php